CLINICAL TRIAL: NCT06062992
Title: Assessing the Optimal Amount of Tissue Sampling in Contrast-Enhanced Stereotactic Biopsy (CESB)
Brief Title: Contrast-Enhanced Stereotactic Biopsy
Acronym: CESB
Status: Recruiting | Type: Observational
Sponsor: Zuyderland Medisch Centrum (Other)
Collaborators: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ZuyderlandMC_CESB
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Cancer Female
Keywords: Breast cancer; Mammography; CEM; Biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Vacuum assisted large core needle biopsies of the breast
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with 'recombined imaging only lesions' or ROLs: Women that recently underwent CEM, which showed a suspicious breast lesion only on the recombined (enhancement) images: a 'recombined image only lesions' or ROL. These women are indicated to undergo CESB.
  Interventions: Diagnostic Test: Contrast Enhanced Stereotactic Biopsy

INTERVENTIONS:
Diagnostic Test: Contrast Enhanced Stereotactic Biopsy — Stereotactic breast biopsy using CEM as targeting modality

SUMMARY:
Contrast-enhanced mammography (CEM) is an emerging breast imaging modality that is based on dual-energy mammography and the injection of iodinated contrast agent. A typical CEM study consists of a low-energy image (equal to a FFDM image) and a recombined image (in which areas of contrast enhancement can be appreciated). However, the situation can occur that lesions are visible only on the recombined (contrast) images (in this protocol defined as 'recombined-only lesions' or ROLs). In these cases, radiologists need to perform 'contrast-enhanced stereotactic biopsy' (CESB), in which CEM is used as a targeting modality.

However, experiences with CESB are still limited and one of the most urgent questions that need to be answered is the amount of tissue sampling that is required to reach a final diagnosis. The investigators aim to study where the cut off will be in terms of tissue sampling volume needed (i.e., number of biopsies) for a reliable diagnosis.

DETAILED DESCRIPTION:
Rationale: Contrast-enhanced mammography (CEM) is an emerging breast imaging modality that is based on dual-energy mammography and the injection of iodinated contrast agent. A typical CEM study consists of a low-energy image (equal to a FFDM image) and a recombined image (in which areas of contrast enhancement can be appreciated). However, the situation can occur that lesions are visible only on the recombined (contrast) images (in this protocol defined as 'recombined-only lesions' or ROLs). In these cases, radiologists need to perform 'contrast-enhanced stereotactic biopsy' (CESB), in which CEM is used as a targeting modality.

However, experiences with CESB are still limited and one of the most urgent questions that need to be answered is the amount of tissue sampling that is required to reach a final diagnosis. The investigators aim to study where the cut off will be in terms of tissue sampling volume needed (i.e., number of biopsies) for a reliable diagnosis.

Objective: To determine the minimum number of CESB-guided tissue samples needed to establish a final histopathological biopsy diagnosis for ROLs.

Study design: Prospective, single center, observational cohort study. Study population: Non-pregnant women (>18 years) able to provide written informed consent and with a ROL recently observed during a regular CEM examination.

Intervention: Included subject will undergo CESB, consisting of an intravenous injection of iodinated contrast agent prior to image acquisition. After administration, a contrast-enhanced stereotactic localization will be performed of the ROL to determine the location and depth of the lesion within the breast. After targeting, 18 samples will be acquired using a 9 Gauge vacuum-assistend biopsy (VAB), collected in six separate and numbered cassettes, to be able to determine the chronological order of the tissue sampling. Each specimen will be histologically analyzed in this chronological order and findings will be compared with the final histopathological result after assessment of all 18 specimens.

Main study parameters/endpoints: The primary study aim will be to calculate the cumulative diagnostic yield per specimen, enabling us to define a minimum number of biopsies required (or tissue volume needed) to establish a reliable diagnosis using CESB. Secondary study outcomes will be general parameters of the biopsy procedure itself, such as patient characteristics, histopathological results, pain experienced during the procedure, and complication rates (hematoma, infection).

ELIGIBILITY:
Inclusion Criteria:

* Women >18 years of age;
* Recent detection of a ROL on CEM;
* Able to provide written informed consent.

Exclusion Criteria:

* All men (male sex);
* Women (female sex) who are contra indicated for CESB (for example: impaired renal function, known hypersensitivity to iodinated contrast);
* Pregnant women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All women recently underwent CEM in our hospital, showing a ROL. Common indications to perform a CEM examination in our hospital are: recalls from breast cancer screening, as problem-solving tool after inconclusive FFDM and/or ultrasound, breast MRI alternative, preoperative staging of breast cancer and baseline examination for women treated with neoadjuvant systemic therapy (where CEM will be used as response monitoring tool).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Amount of tissue needed for CESB | 2 years
  The investigators calculate the diagnostic yield per biopsy sample to establish to minimum amount of tissue samples needed for CESB

SECONDARY OUTCOMES:
Complication rate | 2 years
  The investigators will establish the complication rate of CESB (for example: hematoma, technical failures, infection)
Diagnostic results | 2 years
  The investigators will establish the various diagnostic outcomes (pathology results) of the biopsies performed using CESB
Patient comfort | 2 years
  The investigators will establish the patient (dis)comfort of CESB by scoring the pain associated with this intervention on a 0-10 scale (0 no pain, 10 worst pain ever)

CONTACTS AND LOCATIONS:
Locations (1):
- Zuyderland Medical Center, Sittard, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data can be made available to other researchers.
Supporting Information: Study Protocol, ICF
Time Frame: 2 years
Access Criteria: Signed agreement between institutes